CLINICAL TRIAL: NCT07234188
Title: Comparison of a Procedural Oxygen Mask and High-Flow Nasal Cannula for the Prevention of Hypoxemia During Pediatric Upper Gastrointestinal Endoscopy Under Sedation: A Single-Center Randomized Controlled Pilot Trial
Brief Title: POM vs HFNC for Hypoxemia Prevention in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bedirhan Günel (Other Government)
Responsible Party: Sponsor-Investigator, Bedirhan Günel, Principal Investigator, Kocaeli City Hospital
Organization: Kocaeli City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KSH-ANREA-BG-09
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Experimental): Oxygen delivered via Procedural Oxygen Mask (POM™) at a fixed flow of 15 L/min (approx. FiO₂ 95%) throughout the procedure.
  Interventions: Device: Procedural Oxygen Mask
- Group H (Active Comparator): Oxygen delivered via HFNC at 30 L/min, 35 °C, targeting FiO₂ 95% during the procedure.
  Interventions: Device: High-Flow Nasal Cannula

INTERVENTIONS:
Device: Procedural Oxygen Mask — Delivers oxygen through the mouth and nose during sedation while allowing endoscope passage.
  Arms: Group P
Device: High-Flow Nasal Cannula — Oxygen delivered via HFNC at 30 L/min, 35 °C, targeting FiO₂ 95% during the procedure.
  Arms: Group H

SUMMARY:
Upper gastrointestinal endoscopy is a commonly performed diagnostic and therapeutic procedure in children, allowing evaluation of the esophagus, stomach, and duodenum, as well as interventions such as biopsy, foreign body removal, and polypectomy. Sedation is routinely used, often at greater depths than for standard examinations. Due to anatomical and physiological differences, including smaller airway diameter, higher oxygen consumption, and lower functional residual capacity, pediatric patients are at higher risk of airway obstruction, hypoxemia, and hypoventilation compared to adults. The passage of the endoscope through the mouth further limits airway access and increases the risk of desaturation. Oxygenation during pediatric endoscopy is typically supported using nasal cannulas, high-flow systems, or procedural oxygen masks (POM™). This pilot randomized study aims to compare POM™ and high-flow nasal cannula in preventing hypoxemia during sedated pediatric upper gastrointestinal endoscopy, contributing evidence for safer sedation and airway management practices in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients who consented to participate in the study
* Aged between 6 and 16 years
* Body weight >30 kg
* ASA physical status I-II
* Children scheduled to undergo procedural sedation for non-emergency upper gastrointestinal endoscopy

Exclusion Criteria:

* Lack of parental consent or refusal to sign the participant consent form
* History of endotracheal intubation within the past 3 months
* History of lower respiratory tract infection within the past 3 months
* History of intensive care unit (ICU) admission within the past 3 months
* Presence of a tracheostomy
* History of tracheostomy placement
* Patients with oxygen dependency due to any underlying disease
* Known pulmonary or cardiac disease
* Known congenital craniofacial anomalies
* Congenital or acquired upper airway malformations

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Lowest SpO₂ level during procedure | From the start of sedation to end of endoscopy (typically 5-20 minutes)
  The lowest peripheral oxygen saturation (SpO₂) recorded between the initiation of sedation and the removal of the gastroscope was defined as the primary outcome.
  It was measured via continuous pulse oximetry, and when SpO₂ fluctuated, the value maintained for more than 10 seconds was recorded.

SECONDARY OUTCOMES:
Incidence of hypoxemia | During endoscopic procedure (from sedation start to endoscope removal)
  Defined as any drop in SpO₂ <94% lasting for at least 10 seconds. Based on pulse oximetry recordings.
Number of hypoxemic episodes | During endoscopic procedure
  Recurrent desaturations: counted when SpO₂ falls <94% again, at least 30 seconds after a return to ≥94%.
Duration of hypoxemia (in seconds) | During endoscopic procedure
  Time required for SpO₂ to return to ≥94% after each episode of desaturation (<94%).
Airway interventions | During endoscopic procedure
  Number of occurrences requiring airway maneuvers (chin lift, jaw thrust, or mask ventilation).
Hemodynamic complications | During endoscopic procedure
  Incidence of hypotension (>20% drop from baseline systolic BP), hypertension (>20% increase), bradycardia or tachycardia per age-specific thresholds.
Gastroenterologist satisfaction score | During endoscopic procedure
  Rated from 0 (poor sedation, interrupted) to 10 (optimal sedation).
Incidence of Device Repositioning | During endoscopic procedure
  Adjustment of POM™ or HFNC due to displacement, leakage, or malfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Bedirhan Günel, MD, Principal Investigator — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon reasonable request.